CLINICAL TRIAL: NCT03585907
Title: Feasibility and Efficacy of Dietary Interventions for Older Adults With Subjective Cognitive Decline
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00175761
Record Dates: First submitted 2018-06-21; First posted 2018-07-13 (Actual); Last update posted 2019-10-03 (Actual); Status verified 2019-10

CONDITIONS: Alzheimer Disease; Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Atkins Diet (MAD) (Experimental): A diet that can produce ketones
  Interventions: Dietary Supplement: MAD
- MIND diet (Active Comparator): Mediterranean-DASH Intervention for Neurodegenerative Delay (MIND). A diet that has been indicated to be helpful in preventing or decreasing cognitive decline.
  Interventions: Dietary Supplement: MIND

INTERVENTIONS:
Dietary Supplement: MAD — A high fat, low carbohydrate diet
  Arms: Modified Atkins Diet (MAD)
Dietary Supplement: MIND — A combination of the Mediterranean and DASH diets
  Arms: MIND diet

SUMMARY:
This study aims to assess if/how dietary interventions (i.e., the Modified Atkins Diet (MAD) and/or the Mediterranean-Dietary Approaches to Stop Hypertension (DASH) Intervention for Neurodegenerative Delay (MIND)) might prevent, delay onset, alleviate symptoms, or otherwise alter the course of subjective cognitive decline (SCD) likely due to Alzheimer's disease (AD).

We hypothesize that participants will tolerate both diets well and that the MAD will result in more favorable changes in cognition and other functioning.

DETAILED DESCRIPTION:
Specific aims are to 1) to establish the feasibility of implementing the MAD in older adults with subjective cognitive decline (SCD) likely due to AD, 2) to examine whether changes in participants' cognition, mood, or other functioning are more favorable in patients using the MAD than in patients using the MIND diet, 3) to assess the role of Apolipoprotein E (ApoE) epsilon 4 genotype in response to the MAD in individuals with SCD. We hypothesize that 1) participants will be able to adhere to and tolerate the MAD and the MIND, determined by review of patients' food records and urine ketone production, 2) participants who adhere to the MAD will demonstrate a more favorable change on neuropsychological tests than participants on the MIND diet, and 4) the neuropsychological effects of the MAD will be greatest in those participants without a ε4 allele of the ApoE gene.

ELIGIBILITY:
Inclusion Criteria:

* Self-experienced persistent decline in cognitive capacity compared with a previously normal status that is unrelated to an acute event and that is not explained by a psychiatric disorder or neurological disease apart from Alzheimer's disease, medical disorder, medication, or substance use, with the onset of decline no longer than 5 years prior to study participation
* Clinical Dementia Rating (CDR) score equal to 0
* Montreal Cognitive Assessment (MoCA) equal to or greater than 26
* Age 60 years or older
* Personal physician clearance
* Willing to comply with all requirements of the study protocol and provide informed consent

Exclusion Criteria:

* Diagnosis of mild cognitive impairment (MCI), Alzheimer's disease (AD), or other dementia
* Current psychiatric diagnosis
* Unstable metabolic condition (documented on screening laboratory studies performed within the past year)
* persistent hyponatremia (sodium < 130 mg/dL twice within the past year)
* severe hypernatremia (sodium > 150 mg/dL twice within the past year)
* hypoglycemia (glucose < 50 mg/dL)
* hypocalcemia (albumin-corrected calcium < 8 mg/dL)
* Type-I diabetes
* Type-2 diabetes requiring any medication other than metformin. (Please note that patients with type-2 diabetes may require medication adjustment if on the very low-carb modified Atkins diet.)
* Liver failure
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or ammonia > 5x upper limits of normal
* hyperbilirubinemia
* total bilirubin > 15 mg/dL
* direct bilirubin > 5 mg/dL
* Hypercholesterolemia (on medication, if needed)
* fasting total cholesterol > 300 mg/dL
* fasting LDL cholesterol > 200 mg/dL
* Known fatty acid oxidation disorder or pyruvate carboxylase deficiency
* Body mass index < 18.5
* History of ischemic or hemorrhagic stroke
* History of nephrolithiasis
* History of myocardial infarction or known coronary artery disease
* Acute pancreatitis
* Multiple food allergies or strict dietary requirements
* Any other concerns about nutritional status (e.g., recent unexplained weight loss, difficulty swallowing)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-02 (Estimated); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in Memory Functioning Questionnaire (MFQ) | Baseline/week-0, week-6, completion/week-12
  This is a self-report assessment of cognitive decline. It is rated on a 1-7 scale, with 1 indicating "major problems" and 7 indicating "no problems." It includes 8 sections, each including 1-18 sub-questions. It will be assessed by comparing changes in scores between groups and across time (12 weeks).
Change in Loewenstein-Acevedo Scales of Semantic Interference and Learning (LASSI-L) | Baseline/week-0, week-6, completion/week-12
  This is an assessment of verbal learning and memory for lists of 15 words. More words learned and remembered indicate better learning and memory. It will be assessed by comparing changes in scores between groups and across time (12 weeks).
Change in Para-Rodriguez Short-term Visual Memory Binding Test (SVMBT) | Baseline/week-0, week-6, completion/week-12
  This is an assessment of visual recognition memory for shapes and colors. More accurate recognition indicates better recognition memory. It will be assessed by comparing changes in scores between groups and across time (12 weeks).
Change in Ketone levels | Checked by the participant daily, for 12 weeks/3 months (i.e., from the start day of the diet until the end of the 12 weeks) and checked by the study staff at each study visit (i.e., baseline/week-0, week-3, week-6, and completion/week-12)
  This is detected in urine and measured in mg/dL, with higher levels indicating greater production of ketones and greater adherence to the MAD diet. Adherence will be assessed by percent of participants in the MAD group in at least moderate ketosis (>40 mg/dl) at 3 or more follow-up visits.
MIND Diet Score | 12 weeks/3 months (i.e., from the start day of the diet until the end of the 12 weeks)
  This is assessed by dietitian review of participants daily food logs. Scores range from 0 (not at all adherent) to 15 (perfectly adherent). Any score greater than 9 is considered adherent. It will be assessed by percent of participants in the MIND group with scores of at least 9 at 3 or more follow-up visits.
ApoE epsilon 4 status | Tested via venipuncture or buccal swab at baseline/week-0
  This is a genetic marker of Alzheimer's disease risk. It will be coded as positive (one or more epsilon 4 alleles) or negative (no epsilon 4 alleles). It will be evaluated by stratifying the sample by the presence of at least one ε4 allele and conditioning the efficacy analyses by this variable.

SECONDARY OUTCOMES:
Change in Trail Making Test | Baseline, week-6, week-12
  This is a timed test of processing speed and executive functioning. Faster time to completion and fewer errors indicate better processing speed and executive functioning. It will be assessed by comparing changes in scores between groups and across time (12 weeks).
Change in Prospective Memory Test | Baseline, week-6, week-12
  This is a test of remembering to ask that a borrowed item be returned. The possible scores range from 0 (no cues needed to remember to ask) to 4 (4 cues needed to remember to ask). More cues required indicates worse prospective memory. It will be assessed by comparing changes in scores between groups and across time (12 weeks).
Change in Geriatric Anxiety Scale | Baseline, week-6, week-12
  This is a self-report measure of symptoms of anxiety in older persons. It is rated on a 0 (not at all) to 3 (all of the time) scale. Scores range from 0-90, with higher scores indicating more anxiety. It will be assessed by comparing changes in scores between groups and across time (12 weeks).
Change in Geriatric Depression Scale | Baseline, week-6, week-12
  This is a self-report measure of symptoms of depression in older persons. Items are rated as yes/no. Scores range from 0-30, with higher scores indicating more depression. It will be assessed by comparing changes in scores between groups and across time (12 weeks).

OTHER OUTCOMES:
Change in Cognitive decline concern questionnaire | Baseline, week-6, week-12
  This is a one question questionnaire that asks how concerned/worried a person is about their subjective cognitive decline on a 1 (majorly worried) to 7 (not at all worried) scale, with higher scores indicating a greater degree of concern/worry. It will be assessed by comparing changes in scores between groups and across time (12 weeks).

IPD SHARING:
Plan to Share IPD: Undecided